CLINICAL TRIAL: NCT02031029
Title: A Questionnaire Study by Elevated Prostate Specific Antigen (PSA): Do Men Where Subsequent Assessment Shows Prostate Cancer, Higher Levels of Neuroticism and Stress Compared to Those Who do Not Get the Diagnosis?
Brief Title: Character Traits and Stress in Suspected Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Stopped by the sponsor due to discrepancies in the recruitment process.
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/113
Record Dates: First submitted 2013-10-09; First posted 2014-01-09 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Prostatic Diseases
Keywords: personality scores
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has previously been reported that men with prostate cancer are 1 ) reduced quality of life after diagnosis and treatment, 2 ) neuroticism increases the reduction in QoL related to treatment side effects, and 3) often have very involved and active spouses who seems to have been handed over / taken over parts of the men's responsibility for their own health. We postulate herein a new hypothesis that the stress level is elevated when harbouring undetected prostate cancer. We will investigate whether those who are diagnosed with prostate cancer already in beforehand have an increased degree of masculine stress ( experience of not living up to their own perception of the ideal man ) and neuroticism in the typology. We will examine different personality and QoL questionnaires for patients with elevated PSA, and compare those whose clinical assessment later reveals prostate cancer, with three control groups: 1) men with elevated PSA who are not diagnosed with prostate cancer, 2) men with normal PSA treated for benign prostate enlargement and 3) patient with substantial risk of colorectal cancer (CRC) who undergo colonoscopy, with regard to increased level of masculine stress and the personality trait neuroticism.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Men who are being referred as new urological outpatient and meet the following criteria:

   1. Wanted clinical examined because of elevated PSA
   2. Not strong family history of prostate cancer
   3. It is taken biopsy as part of routine investigation.
2. Control groups: Men being referred to urological / gastroenterological outpatient clinic, and which meet the following criteria:

   1. urination complaints, normal PSA, and study shows prostate size> 40cc
   2. Or melena and cancer suspicion in colorectum
3. Age> 18 years and <75 years

Outcome measures:

Together with statistician look for patterns / covariance in replies from those who are diagnosed with prostate cancer in the questionnaires personality evaluation adapted to normal population (Neo-FFI), gender differentiated stress response questionnaire (MGRSS) and questionnaires related to resilience, relationship and quality of life index, compared with the control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men who be referred a new urological outpatient and satisfy the following:

   * Wanted examined because of elevated PSA
   * Not strong family history of prostate cancer
   * It is taken biopsy as part of routine investigation.
2. Control group: Men referred to urological outpatient clinic, and who satisfy the following

   * urination complaints
   * Normal PSA
   * examination shows prostate size> 40cc
3. Control group: Men first time referred urological / gastroenterological outpatient clinic, and which satisfy the following

   -- symptoms that might indicate cancer suspicion in colorectum
4. Age> 40 years and <75 years

Exclusion criteria:

1. known prostate cancer
2. Reduced consent

4 Familial occurrence of prostate cancer (one or more 1st degree relatives with CaP)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men referred to urological outdoor department or gastroenterological outdoor department
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
MGRSS questionnaire | 2 years
  The profile of the answering patterns will be compared to baseline using psychiatric and statistical evaluation.
Testosterone | 2 years
  Testosterone at baseline and 2 years will be related to wether the patient has confirmed cancer or not.
Cholesterol | 2 years
  Cholesterol at baseline and 2 years will be related to wether the patient has confirmed cancer or not.

SECONDARY OUTCOMES:
Vitamin D, Folic acid, White Blood Cells, C-reactive protein (CRP) | 2 years
  Blood values at baseline and 2 years will be related to wether the patient has confirmed cancer or not.
coffee and green tea consumption | 2 years
  The consumption of coffee and green tea will be related to wether the patient has confirmed cancer or not.

CONTACTS AND LOCATIONS:
Overall Officials: Gunn Iren Meling, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Stavanger University Hospital, urological department, Stavanger

IPD SHARING:
Plan to Share IPD: No